CLINICAL TRIAL: NCT00588900
Title: A Phase II Trial of Irinotecan and AZD2171 in Patients With Metastatic Colorectal Cancer After Progression on First-Line Oxaliplatin, Fluoropyrimidine, and Bevacizumab
Brief Title: Irinotecan and Cediranib in Treating Patients With Metastatic Colorectal Cancer That Did Not Respond to Previous Oxaliplatin, Fluoropyrimidine, and Bevacizumab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-80502; CALGB-80502; CDR0000580967 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2007-12-20; First posted 2008-01-09 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — cediranib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- irinotecan + cediranib (Experimental): Patients receive irinotecan hydrochloride IV over 90 minutes on days 1 and 8 and oral cediranib once daily on days 1-21. Treatment repeats every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.
  After completion of study therapy, patients are followed up every 3 months for up to 2 years from study entry.
  Interventions: Drug: cediranib maleate; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: cediranib maleate
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Cediranib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving irinotecan together with cediranib may kill more tumor cells.

PURPOSE: This phase II clinical trial is studying how well giving irinotecan together with cediranib works in treating patients with metastatic colorectal cancer that did not respond to previous oxaliplatin, fluoropyrimidine, and bevacizumab.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the proportion of patients who are free from progression at 12 weeks from the start of second-line therapy.

Secondary

* To determine objective response rate.
* To determine overall survival.
* To further define the dosing and safety profile of irinotecan hydrochloride and cediranib.

OUTLINE: This is a multicenter study.

Patients receive irinotecan hydrochloride IV over 90 minutes on days 1 and 8 and oral cediranib once daily on days 1-21. Treatment repeats every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for up to 2 years from study entry.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically documented metastatic colorectal cancer

  * The site of the primary lesion must be or have been confirmed endoscopically, surgically, or radiologically to have been in the colon or rectum
  * Patients with a history of histologically proven colorectal cancer treated by surgical resection and who develop radiological or clinical evidence of metastatic cancer do not require additional histological or cytological confirmation of metastatic disease unless either of the following are true:

    * An interval of greater than five years has elapsed between the primary surgery and the development of metastatic disease
    * The primary cancer was stage I
* Must have measurable disease, defined as in at least one dimension (longest dimension to be recorded) as ≥ 20 mm by conventional techniques or as ≥ 10 mm by spiral CT scan

  * Lesions that are considered nonmeasurable include the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* Must have received one and only one prior regimen for metastatic disease containing oxaliplatin, a fluoropyrimidine, and bevacizumab

  * Patients who discontinue oxaliplatin due to toxicity are eligible provided they progressed on the fluoropyrimidine component with or without bevacizumab
* No known brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 8 g/dL
* Leukocytes ≥ 3,000/mm³
* Calculated creatinine clearance > 50 mL/min
* ALT/AST ≤ 2.5 times upper limit of normal (ULN)
* Urine protein < 1+ protein OR protein < 1g by 24-hour urine collection and urine protein:creatinine ratio < 1.0
* Total bilirubin normal
* Not pregnant or nursing
* Negative pregnancy test
* No known end-stage liver disease or active hepatitis
* No colonic or small bowel disorders (e.g., inflammatory bowel disease, Crohn's disease, ulcerative colitis) that predispose to diarrhea in which the symptoms are uncontrolled as indicated by baseline pattern of > 3 watery or soft stools daily in patients without a colostomy or ileostomy

  * Patients with a colostomy or ileostomy may be entered at investigator discretion
* History of hypertension allowed provided it is well controlled (BP < 150/90 mm Hg) on a regimen of antihypertensive therapy
* No concurrent congestive heart failure (New York Heart Association class III or IV)
* No significant history of bleeding events or gastrointestinal (GI) perforation

  * Patients with a history of significant bleeding episodes (e.g., hemoptysis, upper or lower GI bleeding) within 3 months prior to beginning treatment are not eligible unless the source of bleeding has been surgically resected
  * Patients with a history of GI perforation within 12 months prior to beginning treatment are not eligible
* No arterial thrombotic events within 6 months before beginning treatment, including any of the following:

  * Transient ischemic attack
  * Cerebrovascular accident
  * Unstable angina or angina requiring surgical or medical intervention within the past 6 months
  * Myocardial infarction
* No serious or nonhealing wound, ulcer, or bone fracture
* Patients with clinically significant peripheral artery disease (i.e., claudication on ambulating less than one block) or any other arterial thrombotic event within 6 months are also ineligible
* QTc interval ≤ 470 msec
* No personal or family history of long QT syndrome.

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Must have recovered from all acute toxicities of prior therapy for metastatic disease except peripheral neuropathy
* At least 6 weeks between the last dose of bevacizumab and the first dose of cediranib
* Prior pelvic irradiation is allowed (as long as the measurable lesion is outside the radiotherapy field)
* Completed any major surgery ≥ 4 weeks from start of treatment and completed any minor surgery ≥ 1 week prior to start of treatment

  * Insertion of a vascular access device is not considered major or minor surgery from the standpoint of protocol eligibility
  * Patients must have fully recovered from the procedure and have a fully healed incision
* Patients on full-dose anticoagulation (e.g., warfarin) are eligible provided that both of the following criteria are met:

  * The patient has an in-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant or is on a stable dose of low molecular weight heparin
  * The patient has no active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
* Patients receiving anti-platelet agents are eligible
* Patients who are on daily prophylactic aspirin or anticoagulation for atrial fibrillation are eligible
* The use of agents with strong proarrhythmic potential is not permitted during the study
* Patients who received treatment on CALGB-C80405 and whose treatment failed are eligible for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-03; Primary Completion 2010-05 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bert H. O'Neil, MD, Study Chair — UNC Lineberger Comprehensive Cancer Center
Locations (31):
- United States (31):
  - Evanston Hospital, Evanston, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2008 and May 2010, 5 participants were registered.
Groups:
- Irinotecan + Cediranib: Participants receive irinotecan hydrochloride 125 mg/m^2 IV over 90 minutes on days 1 and 8 and oral cediranib 20 mg once daily on days 1-21. Treatment repeats every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Irinotecan + Cediranib
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Irinotecan + Cediranib
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 69.9 [52.3 to 80.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Who Are Progression-free at 12 Weeks From the Start of Second-line Therapy
Description: The 12 week progression-free rate was defined as the percentage of patients that were alive and progression-free 12 weeks after start of second-line therapy. Disease progression was assessed per modified RECIST criteria, and defined as at least a 20% increase in the sum of the longest diameters of target lesions, in either primary or nodal lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of new lesions.
Time Frame: at 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Irinotecan + Cediranib
Number analyzed (Participants) | 5
percentage of participants | 60

2. Secondary Outcome: Radiographic Response Rate
Description: The proportion of patients who respond (completely or partially) to each combination regimen will be estimated.
  Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria: Complete Response (CR): disappearance of all target lesions; Partial Response (PR) 30% decrease in sum of longest diameter of target lesions.
Time Frame: Up to 2 years
Population: Study terminated prematurely; due to patient confidentiality concerns this planned analysis was not performed.
Arm/Group | Irinotecan + Cediranib
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the time from patient randomization to death from any cause. The median OS with 95% CI was estimated using the Kaplan-Meier method.
Time Frame: Up to 2 years
Population: Study terminated prematurely; due to patient confidentiality concerns this planned analysis was not performed.
Arm/Group | Irinotecan + Cediranib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: 4 participants were evaluable for adverse events.
Arm/Group | Irinotecan + Cediranib
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irinotecan + Cediranib (N=4)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
INR increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irinotecan + Cediranib (N=4)
Blood disorder (Blood and lymphatic system disorders) | 2 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (4)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (18)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (7)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 3 (10)
Hepatic pain (Hepatobiliary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 1 (4)
INR increased (Investigations) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (10)
Platelet count decreased (Investigations) | 2 (12)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (4)
Seizure (Nervous system disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (5)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (4)
Thrombosis (Vascular disorders) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less